CLINICAL TRIAL: NCT07224906
Title: Observational Study of the HemoCept Device During Right Heart Catheterization at Boulder Heart
Brief Title: Observational Study of Patients Undergoing Diagnostic Right Heart Catheterization
Status: Recruiting | Type: Observational
Sponsor: HemoCept Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRT-020
Record Dates: First submitted 2025-10-31; First posted 2025-11-05 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Hypertension; Congestive Heart Failure(CHF); Valve Disease, Heart
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this observational pilot study is to collect HemoCept device data from subjects undergoing diagnostic right heart catheterization (RHC) procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects or representatives must have voluntarily signed the informed consent form before any study related procedures.
* Subjects can be any gender but must be age 18 or older.
* Subject is able and willing to provide informed consent and HIPAA authorization.
* Subject is able and willing to meet all study requirements.
* Scheduled for a diagnostic right heart catheterization (RHC-only or combined RHC+LHC; left-heart-only procedures are not eligible)

Exclusion Criteria:

* Subject is pregnant, breastfeeding, or intends to become pregnant during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects above the age of 18 who meet all inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03-06 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Association between device measurements and Pulmonary Capillary Wedge Pressure | Day 1
  The correlation of HemoCept device measurements to Pulmonary Capillary Wedge Pressure (PCWP) measured during right heart catheterization.

CONTACTS AND LOCATIONS:
Locations (1):
- Boulder Heart, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided